CLINICAL TRIAL: NCT05192720
Title: Effect of Supplementary Treatment With Agaricus Blazei Based Mushroom Extract, Andosan, on Patients With Asthma and Allergy
Brief Title: Andosan in Allergic and Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); ImmunoPharma AS (Industry)
Responsible Party: Principal Investigator, Faiza Mahmood, Senior Consultant, Department of Immunology and Transfusion Medicine, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20/01869
Record Dates: First submitted 2021-09-02; First posted 2022-01-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Allergic Asthma; Allergic Rhinoconjunctivitis; Immune Tolerance
Keywords: ASIT; SLIT; Andosan
MeSH Terms: interventions — AndoSan

STUDY DESIGN:
Intervention Model Description: 25-30 patients in each arm receiving Andosan or placebo.
Who Masked: Participant
Masking Description: the patients do not know if they get Andosan or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Andosan (Experimental): The Agaricus blazei Murill-based mushroom extract, Andosan™, is given as one dosage 100 ml/day orally for 1 month. The intervention solution is given in a neutral plastic container
  Interventions: Dietary Supplement: Andosan
- Placebo (Placebo Comparator): The placebo is drinking water with brownish food coloring, given as one dosage 100 ml/day orally for 1 month. The placebo solution is given in a neutral plastic container (same as for intervention/experimental solution).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Andosan — See also detailed study design, Mushroom juice based on Agaricus Blazei and two other types of mushroom.
  Arms: Andosan
Dietary Supplement: Placebo — drinking water with food colour
  Arms: Placebo

SUMMARY:
Examine whether daily oral ingestion of a immunomodulatory mushroom extract (AndoSanTM) in patients with asthma and allergy, undergoing allergen specific immunotherapy experience clinical and biochemical improvement in their disease.

A prospective randomised study comparing the mushroom extract with placebo.

DETAILED DESCRIPTION:
Asthma and allergy are increasing in Norway and Western countries. Treatment is still mostly symptomatic. Extracts of the immunomodulatory and edible mushroom Agaricus blazei, such as Andosan™, have been shown to protect against asthma and allergy in murine models by changing the T helper cell 1(upregulation)-T helper cell 2 (downregulation) balance in the immune system. Positive effects on allergy were also shown in a RCT on blood donors with selfreported allergy. Andosan™ is produced in Japan and approved as food (mushroom juice) in Norway.

The aim of this study is to examine whether Andosan™ i) has similar clinical effects against allergy and asthma in patients as it has in mice, and as earlier shown in a study on blood donors with allergy ii) wether patients taking Andosan has any clinical impact on asthma while taken as supplementary treatment in addition to other medication compared to a placebo group while going through allergen specific immunotherapy (ASIT).

If the extract shows effect on these patients it support the hypotheses that Andosan helps against atopic diseases and facilitate the shift from Th-2 to Th-1 responses at a cellular level.

ELIGIBILITY:
Inclusion Criteria:

* Asthma or allergy patients that are eligible for ASIT (Allergen specific immunotherapy).
* Age above 18.
* Able to understand written and oral Norwegian

Exclusion Criteria:

- none other than not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
FEV1 | 20 days
  Change in FEV1 within-day variation (%) from run-in-period of last five days of intervention.

SECONDARY OUTCOMES:
Oscillometry | 20 days to four weeks
  change in small airway obstruction as measured by the R5Hz and R5-20Hz level in oscillometry.
Questionnaire ACT | four weeks
  Change in asthma symptoms, as measured by the asthma control test
Questionnaire RQLQ | four weeks
  Change in burden of asthma symptoms measured by RQLQ (Respiratory questionnaire of life quality)
Passive basophil cell activation in serum | four weeks
  Difference in activation of basophil cells measured in serum before and after intervention
Immunoglobulin E in serum | four weeks
  difference in concentration before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Mahmood, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus university hospital, Lørenskog, Akershus, Norway